CLINICAL TRIAL: NCT06212609
Title: Optimized and Personalized Trans-cranial Brain Stimulation in Partial Refractory Epilepsies
Acronym: PerEpi2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2021_843_0215
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Transcranial Electric Stimulation; tDCS; Epilepsy; Pharmacoresistant; HR EEG; Children
Keywords: Transcranial electric stimulation; tDCS; Epilepsy; pharmacoresistant; HR EEG; children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transcranial electrical stimulation therapy — new procedure of non-invasive, individualized and optimized transcranial electrical stimulation therapy in the management of pharmaco-resistant focal epilepsies

SUMMARY:
Epilepsy is one of the most common neurological diseases, affecting between 0.5% and 1% of the general population. Therefore, new diagnostic and treatment methods are having a big impact on society. Epilepsy is also one of the most commonly diagnosed pediatric neurological disorders, with long-term implications for the quality of life of those affected and their relatives. In only two-thirds of cases, seizures can be adequately controlled with anticonvulsant drug therapy. For other patients with a drug-resistant focal epilepsy (up to around 2 million in Europe) epilepsy surgery is currently the most effective treatment. However, only 15-20% of these drug-resistant patients are eligible for epilepsy surgery. This is either because the cortical epileptogenic zone cannot be localized with sufficient precision with standard diagnostic means, or because the epileptogenic zone overlaps meaningful cortical areas, so that it cannot be surgically removed without considerable neurological deficit.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, male or female aged 1 to 18, with refractory partial epilepsy considered potentially surgical according to the definition of ILAE. Drug-resistant epilepsy can be defined as the failure of adequate therapeutic trials of two antiepileptics (either monotherapy or in combination) so that the patient is free from seizures on a lasting basis.
* Any epileptic patient with interictal epileptic spikes on his standard or High Resolution EEG and or on the Magnetoencephalography examination
* Any epileptic patient undergoing a structural MRI
* Any patient who has agreed to participate in the PerEpi 1 study allowing the optimization of the location of epileptic sources and the modelling of the optimization of the parameters of transcranial electrical stimulation
* Patients who have at least 4 seizures per month

Exclusion Criteria:

* Patient not meeting the age criteria
* And/or presenting generalized epilepsy
* And/or presenting diffuse interictal peaks and/or presenting a serious alteration of the general condition and vital functions
* And/or in the event of refusal by one of the parents or the child
* Pregnant, parturient or breastfeeding woman.
* Contraindication to the use of mc-tDCS stimulation without seizure

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of remaining seizure number | 10 weeks
  evaluation a new procedure of non-invasive, individualized and optimized transcranial electrical stimulation therapy in the management of pharmaco-resistant focal epilepsies during a study allowing to identify a "proof of concept", in particular for patients who are not eligible for epilepsy surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No